CLINICAL TRIAL: NCT06122142
Title: Advancing Spatial Repellents for Malaria Control: Effectiveness and Cost-Effectiveness of a Spatial Repellent Under Operational Use in Northern Uganda
Brief Title: Spatial Repellents for Malaria Control
Acronym: AEGIS Uganda
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Funder stop request
Sponsor: University of Notre Dame (Other)
Collaborators: S.C. Johnson & Son, Inc. (Industry); Catholic Relief Services (Other); Infectious Diseases Research Collaboration, Uganda (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 23-05-7909
Record Dates: First submitted 2023-10-27; First posted 2023-11-08 (Actual); Last update posted 2025-03-07 (Actual); Status verified 2025-03

CONDITIONS: Malaria
Keywords: Malaria; Spatial Repellent; Transfluthrin; Vector-borne diseases; Mosquito vectors; Incidence
MeSH Terms: conditions — Malaria; Vector Borne Diseases

STUDY DESIGN:
Intervention Model Description: The study design will be a prospective cluster Randomized Control Trial (cRCT)
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Study personnel distribution channel (Active Comparator): SR product will be delivered by paid study personnel.
  Interventions: Device: Transfluthrin - delivery by paid study personnel
- Voucher distribution channel (Experimental): Voucher which will be used to redeem for SR product(s) on a monthly basis for each head of household.
  Interventions: Device: Transfluthrin - delivery by voucher system
- Village health team distribution channel (Experimental): Village health teams will distribute SR products.
  Interventions: Device: Transfluthrin - delivery by village health teams

INTERVENTIONS:
Device: Transfluthrin - delivery by paid study personnel — Passive emanator with formulated transfluthrin, SR product will be delivered by paid study personnel
  Arms: Study personnel distribution channel
Device: Transfluthrin - delivery by voucher system — Passive emanator with formulated transfluthrin, voucher which will be used to redeem for SR product(s) on a monthly basis for each head of household.
  Arms: Voucher distribution channel
Device: Transfluthrin - delivery by village health teams — Passive emanator with formulated transfluthrin, village health teams will distribute SR products.
  Arms: Village health team distribution channel

SUMMARY:
The primary objective of the study is to demonstrate and quantify the effectiveness of a spatial repellent (SR) product, in reducing malaria infection in humans under operational program conditions in a humanitarian assistance context. The design will be a cluster Randomized Control Trial (cRCT) representing an operational research study.

DETAILED DESCRIPTION:
Spatial repellents (SRs) have been widely used for the prevention of mosquito bites, and preliminary findings suggest efficacy against both malaria and Aedes-borne viruses but their effectiveness in reducing mosquito borne diseases under operational use has never been evaluated. SRs have the potential of being critical tools in the prevention of mosquito borne diseases in contexts where typical vectors control strategies, such as Insecticide-Treated Nets (ITNs) and indoor residual spray (IRS), are inaccessible or underutilized such as among displaced peoples or in emergency relief settings. To address this knowledge gap, the Bidibidi refugee settlement in the Yumbe District of North West Uganda was selected as the study site to estimate the impact of the SR on malaria related outcomes under operational use conditions given ongoing humanitarian relief efforts. Children will be enrolled in 3 separate cohorts to establish effectiveness of SRs in reducing malaria infection in distribution channels. One cohort will estimate the direct effect of the SR distributed through a reference channel (study personnel distribution). The two remaining cohorts will estimate the protection of the SR distributed through a voucher channel and village health team (VHT) channel. Cohorts will be followed twice a month (approximately every 15 days) during the first scheduled household visit in the month, a blood sample will be taken for malaria rapid diagnostic test (RDT) (Monthly Visit #1); and, during the second scheduled household visit, a blood sample will only be taken if the participant has a recent history of fever (Monthly Visit #2). The incidence of malaria in each cohort will be estimated and compared to the reference cohort to determine the benefit of using an SR in an area with high, year-round transmission of malaria.

ELIGIBILITY:
Inclusion Criteria:

* Children ≥ 6 months to ≤ 59 months
* Children ≥ 6 months to ≤ 59 months with Hb > 7g/dL and no other serious illness
* Sleeps in cluster (i.e. study area) ≥ 90% of nights during any given month
* Not participating in another clinical trial investigating a vaccine, drug, medical device, or a medical procedure during the Trial
* Provision of informed consent form (ICF) signed by the parent(s) or guardian

Exclusion Criteria:

* Children < 6 months and > 59 months
* Children ≥ 6 months to ≤ 59 months with Hb ≤ 7g/dL with signs of other serious illness or Hb ≤ 7 g/dL with signs of clinical decompensation
* Sleeps in cluster (i.e. study area) < 90% of nights during any given month
* Participating or planned participation in another clinical trial investigating a vaccine, drug, medical device, or a medical procedure during the trial
* No provision of ICF signed by the parent(s) or guardian

Ages: 6 Months to 59 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 0 (Actual)
Dates: Start 2024-05 (Estimated); Primary Completion 2025-05 (Estimated); Study Completion 2025-05 (Estimated)

PRIMARY OUTCOMES:
Effectiveness of SR against malaria infection (both first-time and recurrent). | 12 months
  Measured by rapid diagnostic tests in children aged between 6 months to 59 months.

SECONDARY OUTCOMES:
Cost-effectiveness of SR distribution. | 12 months
  Measure cost of SR implementation in relation to manufacturing, efficacy, and coverage to model projections of cost-effectiveness.
Adverse Events and Serious Adverse Events. | 12 months
  Measured by solicited and unsolicited reports during the intervention period. Mean, minimum and maximum frequency and percentage of Adverse Events and Serious Adverse Eventss across clusters among enrolled subjects will be summarized by distribution channel arm.

CONTACTS AND LOCATIONS:
Overall Officials: John P Grieco, Ph.D., Study Director — University of Notre Dame; Suzanne Van Hulle, M.H.S., Principal Investigator — Catholic Relief Services
Locations (2):
- Uganda (2):
  - Catholic Relief Services, Kampala
  - Infectious Disease Research Collaboration, Kampala

IPD SHARING:
Plan to Share IPD: Yes
Analytical data will be anonymized and GPS tag-blurred to remove sensitive information prior to sharing.
Supporting Information: Study Protocol, SAP, Analytic Code
Time Frame: The data and supporting information will be made available 12 months following completion of data analysis and will remain open access in the public domain.
Access Criteria: Open-access repository distributed under the terms of the Creative Commons Attribution (CC-BY) License, which permits unrestricted use, distribution, and reproduction in any medium, provided the original author and source are credited.

REFERENCES:
- [Background] Achee NL, Bangs MJ, Farlow R, Killeen GF, Lindsay S, Logan JG, Moore SJ, Rowland M, Sweeney K, Torr SJ, Zwiebel LJ, Grieco JP. Spatial repellents: from discovery and development to evidence-based validation. Malar J. 2012 May 14;11:164. doi: 10.1186/1475-2875-11-164. PMID 22583679
- [Background] Hamel MJ, Otieno P, Bayoh N, Kariuki S, Were V, Marwanga D, Laserson KF, Williamson J, Slutsker L, Gimnig J. The combination of indoor residual spraying and insecticide-treated nets provides added protection against malaria compared with insecticide-treated nets alone. Am J Trop Med Hyg. 2011 Dec;85(6):1080-6. doi: 10.4269/ajtmh.2011.10-0684. PMID 22144448
- [Background] Hill N, Zhou HN, Wang P, Guo X, Carneiro I, Moore SJ. A household randomized, controlled trial of the efficacy of 0.03% transfluthrin coils alone and in combination with long-lasting insecticidal nets on the incidence of Plasmodium falciparum and Plasmodium vivax malaria in Western Yunnan Province, China. Malar J. 2014 May 31;13:208. doi: 10.1186/1475-2875-13-208. PMID 24885993
- [Background] Kawada H, Temu EA, Minjas JN, Matsumoto O, Iwasaki T, Takagi M. Field evaluation of spatial repellency of metofluthrin-impregnated plastic strips against Anopheles gambiae complex in Bagamoyo, coastal Tanzania. J Am Mosq Control Assoc. 2008 Sep;24(3):404-9. doi: 10.2987/5743.1. PMID 18939693
- [Background] Lucas JR, Shono Y, Iwasaki T, Ishiwatari T, Spero N, Benzon G. U.S. laboratory and field trials of metofluthrin (SumiOne) emanators for reducing mosquito biting outdoors. J Am Mosq Control Assoc. 2007 Mar;23(1):47-54. doi: 10.2987/8756-971X(2007)23[47:ULAFTO]2.0.CO;2. PMID 17536367
- [Background] Morrison AC, Reiner RC Jr, Elson WH, Astete H, Guevara C, Del Aguila C, Bazan I, Siles C, Barrera P, Kawiecki AB, Barker CM, Vasquez GM, Escobedo-Vargas K, Flores-Mendoza C, Huaman AA, Leguia M, Silva ME, Jenkins SA, Campbell WR, Abente EJ, Hontz RD, Paz-Soldan VA, Grieco JP, Lobo NF, Scott TW, Achee NL. Efficacy of a spatial repellent for control of Aedes-borne virus transmission: A cluster-randomized trial in Iquitos, Peru. Proc Natl Acad Sci U S A. 2022 Jun 28;119(26):e2118283119. doi: 10.1073/pnas.2118283119. Epub 2022 Jun 23. PMID 35737833
- [Background] Ogoma SB, Moore SJ, Maia MF. A systematic review of mosquito coils and passive emanators: defining recommendations for spatial repellency testing methodologies. Parasit Vectors. 2012 Dec 7;5:287. doi: 10.1186/1756-3305-5-287. PMID 23216844
- [Background] Syafruddin D, Asih PBS, Rozi IE, Permana DH, Nur Hidayati AP, Syahrani L, Zubaidah S, Sidik D, Bangs MJ, Bogh C, Liu F, Eugenio EC, Hendrickson J, Burton T, Baird JK, Collins F, Grieco JP, Lobo NF, Achee NL. Efficacy of a Spatial Repellent for Control of Malaria in Indonesia: A Cluster-Randomized Controlled Trial. Am J Trop Med Hyg. 2020 Jul;103(1):344-358. doi: 10.4269/ajtmh.19-0554. Epub 2020 May 14. PMID 32431275
- [Background] The Republic of Uganda Ministry of Health. Annual Health Sector Performance Report Financial Year 2021/22. Ministry of Health, Uganda.
- [Background] Uganda National Malaria Control Division (NMCD), Uganda Bureau of Statistics (UBOS), and ICF. 2019. 2018-19 Uganda Malaria Indicator Survey Atlas of Key Indicators. Kampala, Uganda, and Rockville, Maryland, USA: NMCD, UBOS, and ICF.
- [Background] World Health Organization. Twelfth meeting of the WHO Vector Control Advisory Group. Geneva: World Health Organization; 2020.
- [Derived] Nakyaze E, Van Hulle S, Hembling J, Arinaitwe E, Mbodji M, Alwano MG, Lamwaka FC, Tukwasibwe S, Gonahasa S, Liu F, Grieco JP, Achee NL. Advancing spatial repellents for malaria control: effectiveness and cost-effectiveness of a spatial repellent under operational use in Northern Uganda-study protocol for a cluster randomized controlled trial. Trials. 2024 Aug 22;25(1):555. doi: 10.1186/s13063-024-08378-1. PMID 39175062